CLINICAL TRIAL: NCT04102098
Title: A Phase III, Multicenter, Randomized, Open-Label Study of Atezolizumab (Anti-PD-L1 Antibody) Plus Bevacizumab Versus Active Surveillance as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence After Surgical Resection or Ablation
Brief Title: A Study of Atezolizumab Plus Bevacizumab Versus Active Surveillance as Adjuvant Therapy in Patients With Hepatocellular Carcinoma at High Risk of Recurrence After Surgical Resection or Ablation
Acronym: IMbrave050
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO41535; 2019-002491-14 (EudraCT Number); 2023-504303-86-00 (EU CTIS Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (atezolizumab plus bevacizumab) (Experimental): Participants will receive Atezolizumab + Bevacizumab until disease recurrence or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Arm B (active surveillance) (No Intervention): Active surveillance of participants.

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Arm A (atezolizumab plus bevacizumab)
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 mg/kg on Day 1 of each 21-day cycle.
  Other Names: Avastin
  Arms: Arm A (atezolizumab plus bevacizumab)

SUMMARY:
This study will evaluate the efficacy and safety of adjuvant therapy with atezolizumab plus bevacizumab compared with active surveillance in participants with completely resected or ablated hepatocellular carcinoma (HCC) who are at high risk for disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a first diagnosis of HCC who have undergone either a curative resection or ablation (radiofrequency ablation [RFA] or microwave ablation [MVA] only) within 4-12 weeks prior to randomization
* Documented diagnosis of HCC that has been completely resected or ablated (RFA or MVA only)
* Absence of major macrovascular invasion (except Vp1/Vp2) and extrahepatic spread
* Absence of extrahepatic spread as confirmed by CT or MRI scan of the chest, abdomen, pelvis, and head prior to and following curative procedure
* Full recovery from surgical resection or ablation within 4 weeks prior to randomization
* High risk for HCC recurrence after resection or ablation
* For patients who received post-operative transarterial chemoembolization: full recovery from the procedure within 4 weeks prior to randomization
* For patients with resected HCC, availability of a representative baseline tumor tissue sample
* ECOG Performance Status of 0 or 1
* Child-Pugh Class A status
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Evidence of residual, recurrent, or metastatic disease at randomization
* Clinically significant ascites
* History of hepatic encephalopathy
* Prior bleeding event due to untreated or incompletely treated esophageal and/or gastric varices within 6 months prior to randomization
* Have received more than 1 cycle of adjuvant TACE following surgical resection
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Significant cardiovascular disease within 3 months prior to Day 1 of Cycle 1, unstable arrhythmia, or unstable angina
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Active tuberculosis
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of atezolizumab or within 6 months after the final dose of bevacizumab. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to Day 1 of Cycle 1.
* Co-infection with HBV and HCV
* Co-infection with HBV and hepatitis D viral infection
* Clinical significant uncontrolled or symptomatic hypercalcemia
* Any treatment for HCC prior to resection or ablation, including systemic therapy and locoregional therapy such as TACE
* Treatment with systemic immunostimulatory or immunosuppressive agents
* Inadequately controlled arterial hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease
* Evidence of bleeding diathesis or significant coagulopathy
* Current or recent use of aspirin or full-dose oral or parenteral anticoagulants
* Core biopsy within 3 days of Day 1 of Cycle 1
* History of GI fistula, GI perforation, or intra-abdominal abscess
* Serious non-healing or dehiscing wound
* Major surgical procedure within four weeks
* Chronic daily treatment with a non-steroidal anti-inflammatory drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2027-07-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (134):
- United States (8):
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Mercy Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Inst., Seattle, Washington
- St Vincent's Hospital Sydney, Darlinghurst, New South Wales, Australia
- Austria (3):
  - Lkh-Univ. Klinikum Graz, Graz
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Imeldaziekenhuis, Bonheiden
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (4):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Sociedade beneficente de senhoras Hospital Sirio Libanes, Brasília, Federal District
  - Hospital do Cancer UOPECCAN, Cascavel, Paraná
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- Canada (2):
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- China (36):
  - Anhui Provincial Hospital, Anhui
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Daping Hospital of Third Military Medical University, Chongqing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Cancer Hospital, Fuzhou
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou
  - Cancer Center of Guangzhou Medical University, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Cancer Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Shandong Cancer Hospital, Jinan
  - The 81st Hospital of P.L.A., Nanjing
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - The First Affiliate Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital Fudan Unvierstiy, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - The Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - Northern Jangsu People's Hospital, Yangzhou
- Clinica CIMCA, San José, Costa Rica
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni Thomayerova Nemocnice, Prague
- France (9):
  - Hopital Jean Minoz, Besançon
  - Hôpital Avicenne - Groupement Hospitalier Universitaire Paris Seine St Denis, Bobigny
  - Hôpital Albert Michallon, La Tronche
  - Fondation Hopital Saint Joseph, Marseille
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Hopital Robert Debre, Reims
  - Hopital de Pontchaillou, Rennes
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - Hopitaux de Brabois - Gastro-Entereologie, Vandœuvre-lès-Nancy
- Germany (4):
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik I., Bonn
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt am Main
  - Klinikum der Uni Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Italy (4):
  - Ospedale Regionale Di Parma, Parma, Emilia-Romagna
  - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Azlenda Ospendaliero-Universitaria Pisana, Pisa, Tuscany
- Japan (17):
  - Chiba University Hospital, Chiba
  - Ehime Prefectural Central Hospital, Ehime
  - Hiroshima University Hospital, Hiroshima
  - Sapporo Kosei General Hospital, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Japanese Red Cross Society Himeji Hospital, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Yokohama City University Medical Center, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Osaka Red Cross Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Tokushima University Hospital, Tokushima
  - Toranomon Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Japanese Red Cross Musashino Hospital, Tokyo
- Mexico (2):
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City
- Maastricht University Medical Center, Maastricht, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- Peru (2):
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clínica San Gabriel, Lima
- Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw, Poland
- Russia (4):
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Moscow Oblast
  - Group of companies "Medci", Moskva, Moscow Oblast
  - Clinical hospital #1, FBHI Volga district medical center, Federal Medical and Biological Agency, Nizhny Novgorod, Niznij Novgorod
  - Russian Scientific Center of Radiology and Surgical Technologies, Pesochny, Sankt-Peterburg
- Singapore (2):
  - National Cancer Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (13):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - CHA Bundang Medical Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Boramae Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (3):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital General Universitario Gregorio Marañon, Madrid
- Taiwan (5):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan Uni Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Thailand (4):
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
  - Chulabhorn Hospital, Lak Si
- Adana Baskent University Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Qin S, Chen M, Cheng AL, Kaseb AO, Kudo M, Lee HC, Yopp AC, Zhou J, Wang L, Wen X, Heo J, Tak WY, Nakamura S, Numata K, Uguen T, Hsiehchen D, Cha E, Hack SP, Lian Q, Ma N, Spahn JH, Wang Y, Wu C, Chow PKH; IMbrave050 investigators. Atezolizumab plus bevacizumab versus active surveillance in patients with resected or ablated high-risk hepatocellular carcinoma (IMbrave050): a randomised, open-label, multicentre, phase 3 trial. Lancet. 2023 Nov 18;402(10415):1835-1847. doi: 10.1016/S0140-6736(23)01796-8. Epub 2023 Oct 20. PMID 37871608
- [Derived] Hack SP, Spahn J, Chen M, Cheng AL, Kaseb A, Kudo M, Lee HC, Yopp A, Chow P, Qin S. IMbrave 050: a Phase III trial of atezolizumab plus bevacizumab in high-risk hepatocellular carcinoma after curative resection or ablation. Future Oncol. 2020 May;16(15):975-989. doi: 10.2217/fon-2020-0162. Epub 2020 Apr 30. PMID 32352320

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 134 centers in 26 countries/regions.
Pre-assignment Details: A total of 668 participants were randomized to the Atezo+Bev arm or the Active Surveillance (AS) arm (334 participants in each arm). Participants randomized to the Active Surveillance arm were offered the option to cross over to the Atezo+Bev arm after disease recurrence. 81 participants from the Active Surveillance arm crossed over to receive treatment with Atezo+Bev.
Groups:
- Active Surveillance: Active surveillance of participants.
- Atezolizumab + Bevacizumab: Participants received Atezolizumab + Bevacizumab until disease recurrence or unacceptable toxicity.
Period: Main Study Period
Arm/Group | Active Surveillance | Atezolizumab + Bevacizumab
Started | 334 | 334
Completed | 0 | 0
Not Completed | 334 | 334
Not completed — Ongoing in study | 302 | 291
Not completed — Death | 20 | 27
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 11 | 14
Period: Crossover: AS Who Crossed Over
Arm/Group | Active Surveillance | Atezolizumab + Bevacizumab
Started | 81 | 0
Completed | 0 | 0
Not Completed | 81 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 11 | 0
Not completed — Ongoing in study | 69 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A (Atezolizumab Plus Bevacizumab): Participants received Atezolizumab + Bevacizumab until disease recurrence or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm B (Active Surveillance) | Arm A (Atezolizumab Plus Bevacizumab) | Total
Number analyzed (Participants) | 334 | 334 | 668
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (12.5) | 59.0 (12.1) | 59.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 57 | 113
  Male | 278 | 277 | 555
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 269 | 276 | 545
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 41 | 35 | 76
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival (RFS), as Determined by IRF
Description: RFS is defined as the time from randomization to the first documented occurrence of intrahepatic or extrahepatic HCC as determined by an IRF, or death from any cause (whichever occurs first).
Time Frame: Baseline up to approximately 33 months
Population: The ITT population is defined as all randomized patients, whether or not the patient has received the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B (Active Surveillance) | Arm A (Atezolizumab Plus Bevacizumab)
Number analyzed (Participants) | 334 | 334
Months | NA [21.4 to NA] — Insufficient number of participants with event. | NA [22.1 to NA] — Insufficient number of participants with event.
Statistical Analysis 1: Comparison: Arm B (Active Surveillance) vs Arm A (Atezolizumab Plus Bevacizumab); Stratification factors include geographic region (Asia Pacific excluding Japan vs. rest of world) and High risk features/curative procedure (Ablation vs. Resection with 1 high risk feature vs. Resection with 2 or more high risk features); Test type: Superiority; p = 0.0120, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.93]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

3. Secondary Outcome: RFS as Determined by the Investigator
Description: RFS is defined as the time from randomization to the first documented occurrence of intrahepatic or extrahepatic HCC as determined by an investigator, or death from any cause (whichever occurs first).
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

4. Secondary Outcome: Time to Recurrence (TTR)
Description: TTR defined as the time from randomization to first documented occurrence of intrahepatic or extrahepatic HCC, as determined by the investigator and by an IRF.
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

5. Secondary Outcome: RFS Rate at 24 and 36 Months, as Assessed by the IRF
Time Frame: Randomization up to 24 months and up to 36 months
Reporting Status: Not Posted, anticipated posting 2028-07

6. Secondary Outcome: RFS Rate at 24 and 36 Months, as Assessed by the Investigator
Time Frame: Randomization up to 24 months and up to 36 months
Reporting Status: Not Posted, anticipated posting 2028-07

7. Secondary Outcome: OS Rate at 24 and 36 Months
Description: OS rate defined as the proportion of patients who have not experienced death from any cause at 24 and 36 months after randomization.
Time Frame: Baseline to 24 and 36 months
Reporting Status: Not Posted, anticipated posting 2028-07

8. Secondary Outcome: Time to Extrahepatic Spread (EHS) or Macrovascular Invasion
Description: Time to EHS or macrovascular invasion after randomization, defined as the time from randomization to the first appearance of EHS or macrovascular invasion, as determined by the investigator.
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

9. Secondary Outcome: RFS in Pd-L1-High Subgroup
Description: RFS after randomization as determined by the investigator and by an IRF, among patients in the PD-L1-high subgroup.
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

10. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Baseline up to approximately 91 months
Reporting Status: Not Posted, anticipated posting 2028-07

11. Secondary Outcome: Serum Concentration of Atezolizumab
Description: Serum concentration of atezolizumab.
Time Frame: Prior to any drug administration on Day 1 of Cycles 1, 2, 3, 4, 8, 12, and 16, and 30 minutes after end of atezolizumab infusion on Day 1 of Cycle 1 (each cycle is 21 days)
Population: The pharmacokinetic (PK) analysis population will consist of all patients whom had received any amount of study drug and had at least one measurable serum concentration result post-dose available at the clinical data cutoff for the clinical study report.
Measure: Mean (Standard Deviation); unit: μg/ mL
Arm/Group | Arm A (Atezolizumab Plus Bevacizumab)
Number analyzed (Participants) | 329
μg/ mL
  Cycle 1 Day 1 | NA (NA) — Prior to atezolizumab infusion.
  Cycle 1 Day 1, 30 Min After End of Atezo: number analyzed (Participants) | 310
  Cycle 1 Day 1, 30 Min After End of Atezo | 440 (132)
  Cycle 2 Day 1: number analyzed (Participants) | 317
  Cycle 2 Day 1 | 88.7 (30.4)
  Cycle 3 Day 1: number analyzed (Participants) | 314
  Cycle 3 Day 1 | 137 (53.0)
  Cycle 4 Day 1: number analyzed (Participants) | 305
  Cycle 4 Day 1 | 159 (58.5)
  Cycle 8 Day 1: number analyzed (Participants) | 264
  Cycle 8 Day 1 | 196 (86.2)
  Cycle 12 Day 1: number analyzed (Participants) | 233
  Cycle 12 Day 1 | 202 (90.1)
  Cycle 16 Day 1: number analyzed (Participants) | 192
  Cycle 16 Day 1 | 204 (89.2)

12. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Number of participants with anti-drug antibodies to atezolizumab.
Time Frame: Prior to any drug administration up to approximately 33 month
Population: The immunogenicity analysis population consisted of all participants who received any amount of study drug and had at least one measurable anti-drug antibody (ADA) result post-dose available at the clinical data cutoff for the clinical study report.
Measure: Number; unit: Participants
Arm/Group | Arm A (Atezolizumab Plus Bevacizumab)
Number analyzed (Participants) | 328
Participants
  Baseline evaluable participants | 8
  Post-baseline evaluable participants: number analyzed (Participants) | 324
  Post-baseline evaluable participants | 75

ADVERSE EVENTS:
Time Frame: From the first study drug administration to the data cutoff date: 21 October 2022 (up to approximately 33 months).
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all randomized participants. All-cause mortality reported for the surveillance arm includes participants from the main study period and crossover period. Serious & other adverse events reported based on safety population, which included participants who received any amount of any component of study treatment. Serious and other adverse events were reported separately for participants who crossed over.
Groups:
- Atezolizumab+Bevacizumab: Participants received Atezolizumab + Bevacizumab until disease recurrence or unacceptable toxicity.
- Crossover: Atezolizumab+Bevacizumab: Participants in the Active Surveillance who crossed over to receive Atezo+Bev.
Arm/Group | Active Surveillance | Atezolizumab+Bevacizumab | Crossover: Atezolizumab+Bevacizumab
All-Cause Mortality (participants affected / at risk) | 20/334 | 27/334 | 11/81
Serious Adverse Events (participants affected / at risk) | 34/330 | 80/332 | 10/81
Other Adverse Events (participants affected / at risk) | 111/330 | 296/332 | 63/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance (N=330) | Atezolizumab+Bevacizumab (N=332) | Crossover: Atezolizumab+Bevacizumab (N=81)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 5 (6) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tonsillar neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance (N=330) | Atezolizumab+Bevacizumab (N=332) | Crossover: Atezolizumab+Bevacizumab (N=81)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 12 (12) | 5 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 21 (21) | 4 (5)
Hypothyroidism (Endocrine disorders) | 1 (1) | 47 (49) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 29 (38) | 4 (4)
Fatigue (General disorders) | 4 (4) | 28 (31) | 5 (5)
Oedema peripheral (General disorders) | 2 (2) | 18 (20) | 1 (3)
Pyrexia (General disorders) | 7 (7) | 33 (41) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 25 (27) | 1 (1)
Alanine aminotransferase increased (Investigations) | 18 (19) | 46 (58) | 12 (16)
Aspartate aminotransferase increased (Investigations) | 18 (18) | 51 (67) | 13 (16)
Blood bilirubin increased (Investigations) | 23 (30) | 33 (59) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 17 (26) | 3 (4)
Lymphocyte count decreased (Investigations) | 6 (7) | 22 (37) | 2 (3)
Neutrophil count decreased (Investigations) | 8 (12) | 29 (60) | 5 (5)
Platelet count decreased (Investigations) | 22 (27) | 66 (101) | 17 (19)
Weight increased (Investigations) | 11 (12) | 17 (26) | 0 (0)
White blood cell count decreased (Investigations) | 10 (13) | 28 (76) | 3 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 21 (32) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 40 (43) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 32 (39) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 19 (23) | 2 (3)
Haematuria (Renal and urinary disorders) | 2 (2) | 21 (34) | 3 (3)
Proteinuria (Renal and urinary disorders) | 12 (14) | 153 (227) | 25 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 22 (22) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 20 (23) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 40 (45) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 40 (44) | 9 (9)
Hypertension (Vascular disorders) | 10 (11) | 126 (157) | 25 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04102098/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04102098/SAP_001.pdf